CLINICAL TRIAL: NCT02053025
Title: Appetite Regulation and Mycoprotein
Acronym: mycoprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CRO1332
Record Dates: First submitted 2014-01-22; First posted 2014-02-03 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Appetite; Energy Intake
Keywords: appetite; overweight; energy intake; obesity; gut hormones
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mycoprotein (Active Comparator): 3 levels of mycoprotein will be consumed
  Interventions: Dietary Supplement: mycoprotein
- control protein (Active Comparator): 3 levels of a control protein will be consumed
  Interventions: Dietary Supplement: control protein

INTERVENTIONS:
Dietary Supplement: mycoprotein
  Arms: mycoprotein
Dietary Supplement: control protein
  Arms: control protein

SUMMARY:
The purpose of this study is to investigate the effect of eating various levels of mycoprotein (Quorn) on feelings of appetite, energy intake and levels of gut hormones in overweight volunteers.

DETAILED DESCRIPTION:
Owing to its relatively high protein and fibre content, mycoprotein presents an attractive food product to improve appetite regulation and postprandial glycaemic and insulin responses in overweight and obese individuals at risk of developing T2DM

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 65
* body mass index (BMI) 25-32kg/m2
* Weight stable over the past 6 months
* No known major illness or eating disorder nor on any medication that may impact on appetite or hormone levels.
* No paracetamol or other analgesic in the previous 48 hours
* A score of <2.5 in the Dutch Eating Behaviour Questionnaire (DEBQ)
* A score of <2 in the SCOFF questionnaire

Exclusion Criteria:

* Persons outside the age and BMI ranges stated above
* Pregnant and lactating women
* Weight variation of greater than 5% in the last 6 months
* Any diagnosed major illness
* Any paracetamol or analgesic intake in the last 48 hours
* Diagnosed eating disorder
* Allergy to mycoprotein or mushrooms
* Regular consumption of Quorn products
* Dislike of any of the test foods or drinks
* A score of >2.5 in the Dutch Eating Behaviour questionnaire
* A score of 2 or more in the SCOFF questionaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Energy intake at ad-libitum meal | upon completion of all participants, expected timeframe: 2 years
  Energy intake will be assessed during an ad-libitum meal at 180 minutes at the end of each study visit. Participants will be offered a meal in excess and asked to eat until they feel comfortably full. The meal will be weighed before and after consumption and energy intake will be calculated from the manufacturer's reported nutritional composition.

SECONDARY OUTCOMES:
Glucagon-like peptide-1 (GLP-1) | upon completion of all participants, expected at 2 years
  Plasma glucagon-like peptide-1 (GLP-1) concentrations will be measured by radioimmunoassay (RIA) at the end of the study
peptide tyrosine-tyrosine (PYY) levels | upon completion of all participants, expected at 2 years
  Plasma peptide tyrosine-tyrosine (PYY) concentrations will be measured by radioimmunoassay (RIA) at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NIHR CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bottin JH, Swann JR, Cropp E, Chambers ES, Ford HE, Ghatei MA, Frost GS. Mycoprotein reduces energy intake and postprandial insulin release without altering glucagon-like peptide-1 and peptide tyrosine-tyrosine concentrations in healthy overweight and obese adults: a randomised-controlled trial. Br J Nutr. 2016 Jul;116(2):360-74. doi: 10.1017/S0007114516001872. Epub 2016 May 20. PMID 27198187